CLINICAL TRIAL: NCT00404976
Title: Biomarkers in Exhaled Breath (Condensate) Indicate Presence, Severity and Control of Asthma
Brief Title: Inflammatory Markers in Exhaled Breath (Condensate) in Childhood Asthma
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Other Study IDs: MEC 03-228
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2003-11

CONDITIONS: Asthma; Healthy; Children
Keywords: inflammometry; exhaled breath condensate; fractional exhaled nitric oxide; asthma; children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

Exhaled nitric oxide and inflammatory biomarkers in exhaled breath condensate may be useful to diagnose and monitor childhood asthma. Their ability to indicate an asthma diagnosis, and to assess asthma severity and control, is largely unknown.

Objective:

To study 1) the ability of exhaled nitric oxide and inflammatory markers in exhaled breath condensate (nitrite, nitrate, hydrogen peroxide, 8-isoprostane, interferon-γ, tumor necrosis factor-α, interleukin-2,-4,-5,-10, acidity) to discriminate between childhood asthma and controls. 2) the ability of these biomarkers to indicate asthma severity and control.

Methods:

114 Children were included: 64 asthmatics (10.7±3.0 years, 67.2% atopic) and 50 controls (10.0±0.4 years). Condensate was collected using a glass condenser

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic and control children, aged 5 to 16 years
* Children with doctor-diagnosed asthma, known at the department of Paediatric Pulmonology, University Hospital Maastricht

Exclusion Criteria:

* Presence of a disease that might interfere with the results of this study (e.g. recent upper airway infection, heart disease, anatomic abnormalities of the airways and other chronic inflammatory diseases such as Crohns disease and rheumatoid arthritis)
* Mental retardation
* Inability to perform the EBC procedure properly
* Active smoking
* The use of one of the following medication: Papaverin, Sodium nitroprusside, ACE inhibitors, Oxymetazoline, L-arginine, or NOS inhibitors

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2004-06; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte M Robroeks, MD, Principal Investigator — Maastricht University Medical Center; Edward Dompeling, MD, PhD, Study Director — Maastricht University Medical Center; Quirijn Jöbsis, MD, PhD, Study Director — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands